CLINICAL TRIAL: NCT06907082
Title: Prospective Multicenter Observational Study to Evaluate the Efficacy and Safety of Neoadjuvant Treatment Based on Dual Blockade With Pertuzumab and the Trastuzumab Biosimilar CT-P6 (Herzuma®) in Early HER2-positive Breast Cancer in Routine Clinical Practice
Brief Title: Study to Evaluate the Efficacy and Safety of Neoadjuvant Treatment Based on Dual Blockade With Pertuzumab and the Trastuzumab Biosimilar CT-P6 (Herzuma®) in Early HER2-positive Breast Cancer in Routine Clinical Practice
Acronym: Her-Database
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOCYTIMIB.01
Record Dates: First submitted 2025-03-24; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of pertuzumab and the trastuzumab biosimilar CT-P6 (Herzuma®) in Her2-positive breast ca (Experimental): Combination of pertuzumab and the trastuzumab biosimilar CT-P6 (Herzuma®) in Her2-positive breast cancer susceptible to neoadjuvant chemotherapy.
  Interventions: Drug: Combination of pertuzumab and the trastuzumab biosimilar CT-P6 (Herzuma®) in Her2-positive breast cancer susceptible to neoadjuvant chemotherapy.

INTERVENTIONS:
Drug: Combination of pertuzumab and the trastuzumab biosimilar CT-P6 (Herzuma®) in Her2-positive breast cancer susceptible to neoadjuvant chemotherapy. — Combination of pertuzumab and the trastuzumab biosimilar CT-P6 (Herzuma®) in Her2-positive breast cancer susceptible to neoadjuvant chemotherapy.

SUMMARY:
The study hypothesis is to evaluate whether the pCR rate of neoadjuvant chemotherapy and dual blockade with pertuzumab and the trastuzumab biosimilar CT-P6 (Herzuma®) in HER2-positive early breast cancer in PCH is similar to that reported in clinical trials.

Other aspects to be analyzed include the safety of the combination in PCH, as well as the clinical and tumor characteristics of the study population, assessment of radiological and pathological response, and the role of treatment-induced immunogenicity and the value of plasma HER2 determination.

DETAILED DESCRIPTION:
The study hypothesis is to evaluate whether the pCR rate of neoadjuvant chemotherapy and dual blockade with pertuzumab and the trastuzumab biosimilar CT-P6 (Herzuma®) in HER2-positive early breast cancer in PCH is similar to that reported in clinical trials.

Other aspects to be analyzed include the safety of the combination in PCH, as well as the clinical and tumor characteristics of the study population, assessment of radiological and pathological response, and the role of treatment-induced immunogenicity and the value of plasma HER2 determination.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older.
* Diagnosis of HER2-positive breast cancer confirmed by immunohistochemistry (IHC) of 3+ or positive fluorescence in situ hybridization (FISH) result.
* Early stage without systemic dissemination, amenable to neoadjuvant treatment with chemotherapy and dual anti-HER2 blockade with pertuzumab and the trastuzumab biosimilar CT-P6 (Herzuma®) according to the PCH.

No inclusion staging is established, as the indication will be determined based on standard clinical practice.

* Clinical data available in the patient's medical record for collection.
* Provide written informed consent for the study and informed consent for the Biobank.

Exclusion Criteria:

* Medical or psychiatric incapacity to provide informed consent.
* Known hypersensitivity to trastuzumab or pertuzumab.
* Current treatment with an investigational drug.
* Participation in a clinical trial that involves adding an investigational drug to the standard neoadjuvant clinical treatment with chemotherapy, pertuzumab, and the trastuzumab biosimilar CT-P6 (Herzuma®).
* Withdrawal of consent to participate in the study. The patient may withdraw their consent at any time without having to justify their decision and without any detriment to their clinical care.
* Patient who does not wish to receive or is not a candidate for oncological treatment with chemotherapy or dual anti-Her2 blockade.
* Patient diagnosed with another prognostically relevant neoplastic disease in the previous two years. The exceptions are carcinoma in situ of the cervix or breast, and basal cell or squamous cell carcinoma of the skin.
* Non-neoplastic disease with a prognosis of less than 1 year.
* Medical condition or patient characteristics that, in the investigator's judgment, pose a high risk of serious complications during treatment.
* Being pregnant or breastfeeding.
* Inability to cooperate and comply with the study protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients to be included will be those diagnosed with HER2-positive early breast cancer amenable to neoadjuvant treatment with chemotherapy and dual anti-HER2 blockade.
  Patients will be treated at the hospitals included in the study.
Enrollment: 106 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Up to 18 months
  Pathological complete response (pCR) rate in breast and axillary tissue (ypT0/is ypN0) in patients with HER2-positive early breast cancer after receiving neoadjuvant treatment with chemotherapy, pertuzumab and the trastuzumab biosimilar CT-P6 (Herzuma®) according to routine clinical practice.
  The standard practice for determining pRC is to follow the Miller and Payne criteria. pRC is considered to be grade 5 in tumor tissue, and grade D in the axilla.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Alonso Romero, MD, Principal Investigator — HCUVA
Locations (1):
- HCUVA, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alonso-Romero JL, Martinez-Garcia J, Carrillo-Vicente R, Aramburo AF, Diez AF, Henarejos PS, de la Morena Barrio P, Boix AP, Jimenez MD, Siles JP, Maestre JAP, de Las Heras-Rubio A, Carreno PR. Translational and real-world evidence of trastuzumab biosimilar CT-P6 plus pertuzumab in neoadjuvant HER2-positive early breast cancer. Breast Cancer Res Treat. 2026 Jan 20;215(2):60. doi: 10.1007/s10549-026-07895-8. PMID 41557021